CLINICAL TRIAL: NCT00005644
Title: Phase II Trial of Paclitaxel Plus Gemcitabine in Patients With Advanced Urothelial Carcinoma With Renal Insufficiency
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Cancer of the Urothelium and Decreased Kidney Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067810; E-5899
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; recurrent urethral cancer; distal urethral cancer; proximal urethral cancer; urethral cancer associated with invasive bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Gemcitabine; Paclitaxel

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have advanced cancer of the urothelium with decreased kidney function.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with progressive regional or metastatic transitional cell carcinoma of the urothelium with renal insufficiency when treated with paclitaxel and gemcitabine.
* Determine the toxicity of this regimen in this patient population.

OUTLINE: Patients receive paclitaxel IV over 1 hour followed immediately by gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment continues every 4 weeks for a minimum of 3 courses in the absence of unacceptable toxicity or disease progression.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 10-27 patients will be accrued for this study within 10-27 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed progressive regional or metastatic transitional cell carcinoma of the urothelium

  * Mixed histologies containing a component of transitional cell carcinoma allowed
* Bidimensionally measurable disease
* No clinical evidence of CNS metastases
* Clinically unsuspected organ-confined prostate cancer found at time of cystoprostatectomy allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2.5 times upper limit of normal (ULN) and alkaline phosphatase normal OR
* Alkaline phosphatase no greater than 4 times ULN and SGOT normal OR
* SGOT less than 1.5 times ULN and alkaline phosphatase less than 2.5 times ULN

Renal:

* Creatinine no greater than 3.0 mg/dL
* Glomerular filtration rate no greater than 50 mL/min

Cardiovascular:

* No history of American Heart Association class III or IV heart disease
* No uncontrolled congestive heart failure
* No severe cardiac arrhythmias

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No preexisting peripheral neuropathy grade 2 or greater
* No active unresolved infection requiring parenteral antibiotics within the past 7 days
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior systemic biologic response modifier therapy for advanced disease
* Prior intravesical BCG for superficial disease allowed

Chemotherapy:

* Prior intravesical chemotherapy for superficial disease allowed
* No prior chemotherapy for advanced disease
* At least 6 months since prior adjuvant/neoadjuvant methotrexate, vinblastine, doxorubicin, and cisplatin (MVAC) or cisplatin, methotrexate, and vinblastine (CMV), or cisplatin as a radiosensitizer

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior major surgery and recovered

Other:

* No concurrent hemodialysis

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01-02 (Actual); Primary Completion 2003-02 (Actual); Study Completion 2007-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Vaughn, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (16):
- United States (16):
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - James P. Wilmot Cancer Center, Rochester, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin